CLINICAL TRIAL: NCT01116622
Title: A Phase I Clinical Study of Erlotinib (Tarceva) and Bexarotene (Targretin) Oral Capsules in Advanced Cancers of the Aerodigestive Tract
Brief Title: Erlotinib (Tarceva) and Bexarotene (Targretin) Oral Capsules in Advanced Cancers of the Aerodigestive Tract
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Genentech, Inc. (Industry); Ligand Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0228
Record Dates: First submitted 2010-04-14; First posted 2010-05-05 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2014-11

CONDITIONS: Advanced, Malignant Aerodigestive Tract Tumor (Lung, Head and Neck and Esophagus)
Keywords: Aerodigestive; Targretin; Tarceva
MeSH Terms: interventions — Bexarotene; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daily oral erlotinib and bexarotene capusles (Experimental): Open label dose-ranging trial
  Interventions: Drug: Bexarotene (Targretin®); Drug: Erlotinib (Tarceva™)

INTERVENTIONS:
Drug: Bexarotene (Targretin®) — Level -I 200 mg/m2 Level I 300 mg/m2 Level II 300 mg/m2 Level III 400 mg/m2
  Other Names: Targetin, LGD1069
Drug: Erlotinib (Tarceva™) — Level -1 100mg Level I 100mg Level II 150mg Level III 150mg

SUMMARY:
Primary objective: To determine the Phase II doses and to evaluate the safety of administering bexarotene (Targretin®) daily in combination with oral erlotinib (Tarceva™) to patients with advanced aerodigestive tract cancers.

Secondary objectives: To evaluate the response rates, progression-free survival and overall survival of patients with advanced aerodigestive tract cancers treated with bexarotene (Targretin®) in combination with erlotinib (Tarceva™). To investigate the activity of this targeted combination therapy by evaluating changes in molecular markers from pre- and post-treatment buccal swab samples.

DETAILED DESCRIPTION:
This is a single institution open label dose-ranging trial. Consecutive, eligible patients presenting with the diagnosis of advanced aerodigestive tract malignancy are to be enrolled in this study. All eligible patients will receive continuous daily oral erlotinib (Tarceva™) with daily bexarotene oral capsules (Targretin®). The two agents will be taken at the same time. Three dose levels of daily bexarotene in combination with daily erlotinib will be studied.

Eligible patients will be entered in cohorts of three at each dose level. Doses will not be escalated over the course of treatment of an individual patient. If a single patient experiences grade 4 hematologic or ≥ grade 3 non-hematologic toxicity (excluding hyperlipidemia and nausea/vomiting), the next group of three patients will be entered at the same dose. A maximum of 6 evaluable patients will be enrolled at any one dose level. Dose escalation is performed after all patients (3 or 6) at the previous dose level have received treatment for 4 weeks. Treatment will continue until progression of disease, unacceptable adverse effects, or patient refusal. If grade 4 hematologic or ≥ grade 3 non-hematologic toxicity (excluding hyperlipidemia and nausea/vomiting) is observed in two or more patients on dose level 1, the next three patients (or six if similar toxicity develops in one of the first three patients) will receive dose level -1. If such toxicity is seen in two or more patients, the trial will be terminated. We anticipate the maximum accrual of 18 patients to this trial.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmation of advanced malignant aerodigestive tract tumo(lung, head and neck and esophagus)
* No known curative treatment.
* Age >18 years
* Karnofsky performance status ≥ 60%.
* Prior chemotherapy or radiotherapy is allowed.
* Fasting triglycerides equal or less than upper limit of normal
* Female patients and male patients with female partners of childbearing potential must agree to sexual abstinence or to practice effective contraception (recommended to be two reliable forms of non-hormonal contraception used simultaneously) during the entire period of Targretin capsule treatment and for at least one (1) month after treatment is discontinued. Male patients with female sexual partners who are pregnant, or possibly pregnant or who could become pregnant during the study must agree to use condoms during sexual intercourse during the entire period of Targretin capsule treatment and for at least one (1) month after the last dose of Targretin capsules.
* All patients must give informed consent indicating they are aware of the investigational nature of this treatment.

Exclusion Criteria:

* Organ dysfunction that precludes use of bexarotene or erlotinib:
* hepatic dysfunction, as evidenced by either:

  * transaminase (SGOT or SGPT) > 2.5 X upper limit of normal (ULN) or > 5 X ULN if known liver metastases
  * bilirubin > upper limit of normal
* renal dysfunction, as evidenced by calculated creatinine clearance < 30 ml/min
* A serious uncontrolled medical disorder or active infection which would impair their ability to receive study treatment will be excluded.
* Significant cardiac disease, including uncontrolled high blood pressure, unstable angina, congestive heart failure, myocardial infarction within the previous 3 months or serious cardiac arrhythmias will be excluded. Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol will be excluded.
* Concurrent use of other anti-cancer investigational agents is not allowed
* Women who are pregnant or breast-feeding and women of childbearing potential or fertile males not using an adequate method of birth control will be excluded.
* Known hypersensitivity to bexarotene, erlotinib or other components of the capsules.
* Risk factor for pancreatitis (e.g., prior pancreatitis, uncontrolled hyperlipidemia,excessive alcohol consumption, uncontrolled diabetes mellitus, biliary tract 10 disease, and medications known to increase triglyceride levels or to be associated with pancreatic toxicity).
* Systemic anticancer therapy of any kind within 14 days prior to initiating study medications.
* Investigational therapy of any kind within 30 days prior to initiating study medications.
* Systemic vitamin A in doses exceeding 15,000 IU/day within 14 days prior to initiating study medications.
* Unwillingness or inability to minimize exposure to sunlight and artificial ultraviolet light while receiving the capsules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Phase II dose determination and evaluation of the safety of administering bexarotene(Targretin®) daily in combination with oral erlotinib (Tarceva™) to patients with advanced aerodigestive tract cancers. | When final patient is removed from study or at the discreation of the investigator
  The purpose of this study is to evaluate the safety of daily oral administration of bexarotene in combination with erlotinib at three dose levels to patients with advanced aerodigestive tract cancer. At least 3 patients will be entered onto each dose level. Dose limiting toxicity is defined as grade 3 or greater non-hematologic toxicity or grade 4 hematologic toxicity. The recommended Phase II dose is defined as the highest dose level of bexarotene oral capsules in combination with oral erlotinib that induces DLT in fewer than 33% of patients.

SECONDARY OUTCOMES:
Response rates, progression-free survival and overall survival of patients with advanced aerodigestive | When final patient is removed from study or at the discretion of the investigator
  Response rates will be described using RECIST criteria wherever possible. Survival will be determined by the number of days from study entry until death or date of last known followup and will be analyzed using the Kaplan-Meier method. Time to progression is defined as the interval from the initiation of treatment to the occurrence of progression or to last contact, or to the start of other antitumor therapy.
Investigate the activity of this targeted combination therapy by evaluating changes in molecular markers from pre- and post-treatment buccal swab samples. | When final patient is removed from study or at the discretion of the investigator

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin H. Dragnev, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States